CLINICAL TRIAL: NCT01203514
Title: The Effects of Erythropoietin (EPO) on the Transfusion Requirements of Preterm Infants 401-1250 Grams: Two Multi-Center, Randomized, Double-Masked, Placebo Controlled Studies
Brief Title: The Effects of Erythropoietin (EPO) on the Transfusion Requirements of Very Low Birth Weight Infants
Acronym: EPO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Robin K. Ohls, Lead Principal Investigator, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0017; U10HD027853 (NIH); M01RR008084 (NIH); U10HD027851 (NIH); M01RR000039 (NIH); U10HD034167 (NIH); M01RR002635 (NIH); M01RR002172 (NIH); M01RR001032 (NIH); U10HD027856 (NIH); M01RR000750 (NIH); U10HD027881 (NIH); M01RR000997 (NIH); U10HD021415 (NIH); U10HD021385 (NIH); U10HD027871 (NIH); M01RR006022 (NIH)
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Anemia, Neonatal
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Prematurity; Erythrocyte transfusions; Erythropoietin (Epo); Blood loss; Phlebotomy
MeSH Terms: conditions — Premature Birth; Anemia, Neonatal; Hemorrhage | interventions — Erythropoietin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Trial 1 Experimental (Experimental): Infants 401-1,000g birthweight
  Interventions: Drug: Erythropoietin
- Trial 1: Sham Comparator (Sham Comparator): Infants 401-1,000g birthweight
  Interventions: Other: Sham Comparator
- Trial 2: Experimental (Experimental): Infants 1,001-1,250g birth weight
  Interventions: Drug: Erythropoietin
- Trial 2: Sham Comparator (Sham Comparator): Infants 1,001-1,250g birth weight
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Drug: Erythropoietin — Infants received 400 U/kg Erythropoietin (Epo) 3 times weekly and a weekly intravenous infusion of 5 mg/kg iron dextran until they had an enteral intake of 60 mL/kg/d.
  Other Names: Human recombinant erythropoietin
  Arms: Trial 1 Experimental; Trial 2: Experimental
Other: Sham Comparator — Infants in the placebo/control group received sham subcutaneous injections when intravenous access was not available.
  Arms: Trial 1: Sham Comparator; Trial 2: Sham Comparator

SUMMARY:
This study tested the safety and efficacy of transfusing erythropoietin (Epo) and iron in infants of <1,250g birth weight. For infants 401-1,000g birth weight, we tested whether early erythropoietin (Epo) and iron therapy would decrease the number of transfusions received. For infants 1,001-1,250g birth weight, we tested whether early erythropoietin (Epo) and iron therapy would decrease the percentage of infants who received any transfusions.

DETAILED DESCRIPTION:
Critically ill preterm infants experience in the first 1-2 weeks after birth daily blood losses that may equal 5-10% of their total blood volume. Such losses and associated anemia typically result in multiple erythrocyte transfusions. This iatrogenic anemia commonly is followed by the anemia of prematurity, prompting additional transfusions.

This study tested the safety and efficacy of transfusing erythropoietin (Epo) and iron in infants of <1,250g birth weight. For infants 401-1,000g birth weight (Trial 1), we tested whether early erythropoietin (Epo) and iron therapy would decrease the number of transfusions received. For infants 1,001-1,250g birth weight (Trial 2), we tested whether early erythropoietin (Epo) and iron therapy would decrease the percentage of infants who received any transfusions.

Therapy was initiated by day of life 4 and continued through the 35th postmenstrual week. Infants were randomized to receive either Epo and iron therapy or a sham procedure. Treated infants received 400 U/kg Epo 3 times weekly and a weekly intravenous infusion of 5 mg/kg iron dextran until they had an enteral intake of 60 mL/kg/d. Infants in the placebo/control group received sham subcutaneous injections when intravenous access was not available. Complete blood and reticulocyte counts were measured weekly, and ferritin concentrations were measured monthly.

Transfusions were administered according to protocol. Infants did not receive a transfusion solely to replace blood lost through phlebotomy. Infants who met transfusion criteria received a transfusion of 15 mL/kg packed red blood cells (PRBC) for a hematocrit of >25% or 20 mL/kg PRBC for a hematocrit of <=25%. Blood losses and transfusion data were recorded.

Trial 2 was terminated after enrollment of 118 infants after the Data and Safety Monitoring Committee reviewed the final results of Trial 1 and preliminary results of Trial 2. On the basis of these data, the Committee concluded that it was statistically unlikely that Trial 2 would demonstrate a significant decrease in the percentage of infants who would receive a transfusion during the study.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a birth weight of 4010-1250g, <32 weeks' gestation, and 24-96 hours old at the time of study entry
* Likely to survive >72 hours
* Informed consent from a parent or guardian.

Exclusion Criteria:

* Major congenital anomaly
* A positive direct antiglobulin test
* Evidence of coagulopathy
* Clinical seizures
* Systolic blood pressure >100 mm Hg (in the absence of pressor support)
* Absolute neutrophil count (ANC) of <=500/micro-L

Ages: 24 Hours to 96 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 318 (Actual)
Dates: Start 1997-08; Primary Completion 1998-08 (Actual); Study Completion 2000-08 (Actual)

PRIMARY OUTCOMES:
Erythrocyte transfusions in infants 401-1,000g birthweight | Hospital discharge or 35 weeks postmenstrual age
Blood transfusions | Hospital discharge or 35 weeks postmenstrual age

CONTACTS AND LOCATIONS:
Overall Officials: Robin K. Ohls, MD, Study Director — University of New Mexico; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Barbara J. Stoll, MD, Principal Investigator — Emory University; Ann R. Stark, MD, Principal Investigator — Brigham and Women's Hospital; James A. Lemons, MD, Principal Investigator — Indiana University; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Study Director — Yale University; Raymond Bain, PhD, Principal Investigator — George Washington University
Locations (9):
- United States (9):
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Harvard University, Cambridge, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - University of Tennessee, Memphis, Tennessee

REFERENCES:
- [Result] Ohls RK, Ehrenkranz RA, Wright LL, Lemons JA, Korones SB, Stoll BJ, Stark AR, Shankaran S, Donovan EF, Close NC, Das A. Effects of early erythropoietin therapy on the transfusion requirements of preterm infants below 1250 grams birth weight: a multicenter, randomized, controlled trial. Pediatrics. 2001 Oct;108(4):934-42. doi: 10.1542/peds.108.4.934. PMID 11581447
- [Result] Ohls RK, Ehrenkranz RA, Das A, Dusick AM, Yolton K, Romano E, Delaney-Black V, Papile LA, Simon NP, Steichen JJ, Lee KG; National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental outcome and growth at 18 to 22 months' corrected age in extremely low birth weight infants treated with early erythropoietin and iron. Pediatrics. 2004 Nov;114(5):1287-91. doi: 10.1542/peds.2003-1129-L. PMID 15520109
- See also: NICHD Neonatal Research Network — http://neonatal.rti.org/